CLINICAL TRIAL: NCT02005926
Title: Phase II Trail of Removing Sonographic Abnormal Lymph Node in Sentinel Lymph Node Biopsy of Breast Cancer Patient
Brief Title: The Accuracy of Sentinel Node Biopsy of Breast Cancer With Sonographic Abnormal Axillary Lymph Nodes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tao OUYANG (Other)
Responsible Party: Sponsor-Investigator, Tao OUYANG, Chairman of Breast Center, Peking University
Organization: Peking University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BCP07
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Sentinel lymph node biopsy; Ultrasonography; Fine needle aspiration
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- negative FNA result of abnormal node (Experimental): Axillary ultrasound examination was undergone for all breast cancer patients before sentinel lymph node biopsy (SLNB). If abnormal axillary lymph node was found, ultrasound-guided FNA cytology of these nodes were performed. The abnormal nodes were defined as completely hypoechoic node, asymmetric focal hypoechoic node, cortical lobulation and cortical thickness >3mm. Patients with negative results of FNA would undergo SLNB. Technetium-99m-labeled Rituximab was used for lymphatic mapping. Before the SLNB operation, a hookwire was placed at the suspicious axillary lymph node by ultrasound guidance. In the SLNB operation, radioactive nodes and wire-localized nodes were removed and labeled separately for pathological examination.
  Interventions: Procedure: Wire-localized abnormal node

INTERVENTIONS:
Procedure: Wire-localized abnormal node — Before the sentinel lymph node biopsy (SLNB) operation, a hookwire was placed at the suspicious axillary lymph node by ultrasound guidance to localize the abnormal node. In the SLNB operation, radioactive nodes and wire-localized nodes were removed and labeled separately for pathological examination.

SUMMARY:
* This is a phase II, prospective, single-center, non-randomized, non-controlled study.
* Sentinel lymph node biopsy (SNB) is a standard staging procedure in early breast cancer. The potentially increasing false negative rate of SNB was concerned if the sonographic abnormal node was not excised. The aim of this study was to evaluate the accuracy of SNB in breast cancer with sonographic abnormal axillary lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmsed primary breast cancer by core neelde biopsy or excisional biospy
* abnormal axillary lymph node was found by ultrasound examination before SLNB (abnormal nodes were defined as completely hypoechoic node, asymmetric focal hypoechoic node, cortical lobulation and cortical thickness >3mm)
* ultrasound-guided FNA cytology of these nodes were performed
* the result of FNA cytology was negative (no tumour cell was found)
* patient planed to perform SLNB

Exclusion Criteria:

* pathological diagnosed ductal carcinoma in situ by excisional biospy
* abnormal axillary lymph node was found by ultrasound examination but FNA cytology of these nodes were not performed
* the result of FNA cytology was positive (tumour cell was found)
* T4d tumour
* patient has recieved neo-adjuvant system therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-05; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
False negative rate of sentinel node biopsy if sonographic abnormal node not be removed | one week after sentinel node biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoqing Fan, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Breast cancer, Peking University Cancer Hospital & Institute, Beijing, China